CLINICAL TRIAL: NCT06325631
Title: Comparative Evaluation of the Results of Facet Joint Injections Performed by Using Fluoroscopy, Ultrasound Guidance and Anatomic Location Administered to the Patients With Facet Syndrome
Brief Title: Comparative Evaluation of the Results of Facet Joint Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oznur Uzun (Other)
Responsible Party: Sponsor-Investigator, Oznur Uzun, Principal Investigator, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Ankara City Hospital Bilkent
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain, Mechanical; Facet Syndrome of Lumbar Spine
Keywords: facet joint syndrome; low back pain; fluoroscopy; ultrasound
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluoroscopy (Experimental)
  Interventions: Procedure: Intra-articular injection to lumbar facet joint
- Ultrasound (Experimental)
  Interventions: Procedure: Intra-articular injection to lumbar facet joint
- Anatomic (Experimental)
  Interventions: Procedure: Intra-articular injection to lumbar facet joint

INTERVENTIONS:
Procedure: Intra-articular injection to lumbar facet joint — to treat low back pain caused by facet joint syndrome

SUMMARY:
Low back pain affects 60 to 90% of the total population. It is one of the most common causes of disability in adults. Low back pain can be originated from a wide variety of structures, and the facet joint is one of these structures. It is thought that 21 to 41% of low back pain originates from the facet joint. A wide variety of conservative treatments, including intra-articular injections, are used to treat low back pain originating from the facet joint. However, there is still no consensus on the most effective treatment method. With appropriate patient selection, facet joint injections can provide significant improvements in patients' pain scores. After Goldthwait defined the facet joint concept in 1911, Ghormley defined facet joint syndrome in 1933. The source of pain in 40-50% of patients is the lumbar facet joints. Innervation of the lumbar facet joints is provided by the medial branches of the dorsal roots of the spinal nerves. In 1975, Shealy described the coagulation of the articular nerve support of the spinal facet joints with the radiofrequency method. These methods have been further developed over time. The results of facet joint injections are satisfactory in well-selected patient groups. It has been shown that intra-articular steroid injection to the facet joint is superior to systemic steroid use in patients with low back pain. In this study, it was aimed to methodically compare the facet joint injections applied to patients diagnosed with facet syndrome in the outpatient clinic of the Physical Therapy and Rehabilitation Hospital in terms of patient pain scores, application time, effort spent and patient anxiety. Intra-articular injections will be performed under by fluoroscopy or ultrasound guidance or anatomic location.

ELIGIBILITY:
Inclusion Criteria:

* Patients with facet joint syndrome diagnosis

Exclusion Criteria:

* pregnant patients
* breastfeeding patients
* patients with cardiac pacemaker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | VAS will be applied to the patients before the procedure and at the first and twelfth week after the procedure
  Pain intensity will be measured with Visual Analogue Scale, which is used to measure musculoskeletal pain with very good reliability and validity. Visual Analogue Scale is between 0-10 cm. 0 means no pain, 10 means the most severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomez Vega JC, Acevedo-Gonzalez JC. Clinical diagnosis scale for pain lumbar of facet origin: systematic review of literature and pilot study. Neurocirugia (Engl Ed). 2019 May-Jun;30(3):133-143. doi: 10.1016/j.neucir.2018.05.004. Epub 2018 Jun 14. English, Spanish. PMID 29910103
- [Result] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Evaluation of lumbar facet joint nerve blocks in managing chronic low back pain: a randomized, double-blind, controlled trial with a 2-year follow-up. Int J Med Sci. 2010 May 28;7(3):124-35. doi: 10.7150/ijms.7.124. PMID 20567613
- [Result] Nelson AM, Nagpal G. Interventional Approaches to Low Back Pain. Clin Spine Surg. 2018 Jun;31(5):188-196. doi: 10.1097/BSD.0000000000000542. PMID 28486278
- [Result] Baroncini A, Maffulli N, Eschweiler J, Knobe M, Tingart M, Migliorini F. Management of facet joints osteoarthritis associated with chronic low back pain: A systematic review. Surgeon. 2021 Dec;19(6):e512-e518. doi: 10.1016/j.surge.2020.12.004. Epub 2021 Feb 10. PMID 33582054